CLINICAL TRIAL: NCT02885649
Title: Pilot Study of the Blockade of Androgens in Renal Cell Carcinoma Using Enzalutamide (BARE)
Brief Title: Enzalutamide Before Surgery in Treating Patients With Kidney Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric A. Singer, MD, MA, MS, FACS, Principal Investigator, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro20170000806; NCI-2016-01113 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 081604 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Clear Cell Renal Cell Carcinoma; Stage I Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — enzalutamide; Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzalutamide, nephrectomy) (Experimental): Patients receive enzalutamide PO daily for 90 days in the absence of disease progression or unacceptable toxicity. Patients then undergo partial or radical nephrectomy.
  Interventions: Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Procedure: Nephrectomy

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Nephrectomy — Undergo partial or radical nephrectomy

SUMMARY:
This pilot phase 0 trial studies how well enzalutamide works before surgery in treating patients with kidney cancer. Androgens are a type of hormone produced by the body that may cause kidney tumors to grow. Anti-hormone therapy, such as enzalutamide, may lessen the amount of androgens produced by the body and keep kidney tumors from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the effects of neoadjuvant enzalutamide on clear cell renal cell carcinoma (ccRCC).

OUTLINE:

Patients receive enzalutamide orally (PO) daily for 90 days in the absence of disease progression or unacceptable toxicity. Patients then undergo partial or radical nephrectomy.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical T1N0M0 (=< 7 cm) renal mass as measured on cross-sectional imaging (computed tomography [CT] or magnetic resonance imaging [MRI])
* Biopsy proven ccRCC
* Tumor with androgen receptor (AR) expressed >= 4580 copies/ug ribonucleic acid (RNA)
* Can provide informed consent
* Adequate hepatic function (>= 1.5 x upper limit of normal [ULN]; patient's with Gilbert's disease are not excluded)
* Adequate renal function (estimated glomerular filtration rate [GFR] > 40mL/min)
* No evidence of metastatic disease on baseline imaging (chest x-ray [CXR] or chest CT, abdominal CT or MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2

Exclusion Criteria:

* Prior use of androgen deprivation including enzalutamide
* Pregnant women or women who are of child bearing age who are not willing to use two (2) forms of contraception during treatment with enzalutamide and for six (6) months after treatment
* Men must use adequate methods of contraception during and at least 3 months after treatment if engaging in sexual activity with a female of child bearing age
* Known hypersensitivity to enzalutamide
* History of unprovoked deep vein thrombosis/pulmonary embolism (DVT/PE) in past twelve (12) months
* Inability to stop anticoagulants/antiplatelet therapy peri-operatively
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma)
* History of loss of consciousness or transient ischemic attack within twelve (12) months of enrollment
* Any unstable, serious co-existing medical conditions including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within twelve (12) months prior to screening
* Known or suspected brain metastasis or active leptomeningeal disease
* Current use of exogenous testosterone
* Retroperitoneal/hilar adenopathy concerning for locally advanced disease
* Metastatic RCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Cell proliferation | Up to 36 months
Tumor apoptosis as measured by annexin | Up to 36 months

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) as assessed by Common Terminology Criteria for Adverse Events version 4 | Up to 36 months
  Post-operative complications will be documented according to the Clavien-Dindo Classification System.
Tumor size as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 36 months

OTHER OUTCOMES:
AR expression measured in pre- and post-treatment tissue samples by immunohistochemistry (IHC) | Up to 36 months
  Pre- and post-treatment ccRCC samples will be used to purify mRNA, construct cDNA, and perform qPCR to quantify expression of mRNA. IHC staining will be performed on ccRCC pre- and post-treatment.
Genome-wide analysis of post-treatment tissue samples assessed by whole exome and RNA sequencing | Up to 36 months
Intracrine androgen signaling levels of testosterone and dihydrotestosterone assessed in tissue | Up to 36 months
  Pre- and post-treatment tissue levels of testosterone and dihydrotestosterone will be compared to their respective serum levels to assess intracrine androgen signaling in ccRCC following enzalutamide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Singer, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States